CLINICAL TRIAL: NCT01193907
Title: A Phase 2, Randomized, Observer-blind, Controlled, Single Center Study to Evaluate the Safety and Immunogenicity of Three Formulations of the Novartis Vaccines Institute for Global Health (NVGH) Glycoconjugate Vaccine Against S. Typhi in Adult Subjects 18 to 40 Years of Age
Brief Title: Safety and Immunogenicity of Three Formulations of Vi-CRM197 Vaccine Against S. Typhi in Adults (18-40 Years Old)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H01_04TP; 2010-021874-12 (EudraCT Number)
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Typhoid Fever
Keywords: Typhoid fever; Glycoconjugate vaccine; Vi polysaccharide; Immunogenicity
MeSH Terms: conditions — Typhoid Fever | interventions — Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- NVGH Vi-CRM197 conjugate vaccine 12.5 mcg (Experimental): 1 dose of 0.5 mL containing 12.5 mcg of Vi-CRM
  Interventions: Biological: NVGH Vi-CRM197 12.5 mcg
- NVGH Vi-CRM197 conjugate vaccine 5 mcg (Experimental): 1 dose of 0.5 mL containing 5 mcg of Vi-CRM
  Interventions: Biological: NVGH Vi-CRM197 5.0 mcg
- NVGH Vi-CRM197 conjugate vaccine 1.25 mcg (Experimental): 1 dose of 0.5 mL containing 1.25 mcg of Vi-CRM
  Interventions: Biological: NVGH Vi-CRM197 1.25 mcg
- Typherix (Active Comparator): 1 dose of 0.5 mL containing 25 mcg of Vi-polysaccharide
  Interventions: Biological: Vi-polysaccharide vaccine

INTERVENTIONS:
Biological: NVGH Vi-CRM197 12.5 mcg — 1 dose of 0.5 mL
  Arms: NVGH Vi-CRM197 conjugate vaccine 12.5 mcg
Biological: NVGH Vi-CRM197 5.0 mcg — 1 dose of 0.5 mL
  Arms: NVGH Vi-CRM197 conjugate vaccine 5 mcg
Biological: NVGH Vi-CRM197 1.25 mcg — 1 dose of 0.5 mL
  Arms: NVGH Vi-CRM197 conjugate vaccine 1.25 mcg
Biological: Vi-polysaccharide vaccine — 1 dose of 0.5 mL containing 25 mcg of Vi polysaccharide
  Arms: Typherix

SUMMARY:
This trial is aimed to evaluate the safety and immunogenicity profiles of three formulations of Vi-CRM197 conjugate vaccine against S. Typhi in healthy human adults in comparison with the currently licensed Vi polysaccharide vaccine

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of age ≥18 to ≤40 years.
2. Individuals who, after the nature of the study have been explained to them, have given written consent according to local regulatory requirements.
3. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.
4. Individuals with negative urine screening tests for drug addition (Opiate, Cocaine, Amph/Metamphetamine, Cannabinoides )
5. If women, use of birth control one month before study start, a negative pregnancy test and willingness to use birth control measures for the entire study duration.

Exclusion Criteria:

1. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
2. Individuals with any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
3. Individuals who are not able to understand and to follow all required study procedures for the whole period of the study.
4. Individuals with history of any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
5. Individuals with known or suspected HIV infection or HIV related disease, with history of an autoimmune disorder or any other known or suspected impairment /alteration of the immune system, or under immunosuppressive therapy including use of systemic corticosteroids or chronic use of inhaled high-potency corticosteroids within the previous 30 days, or were in chemotherapy treatment within the past 6 months.
6. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
7. Individuals with any serious chronic or progressive disease according to judgment of the investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
8. Individuals who have any malignancy or lymphoproliferative disorder.
9. Individuals with history of allergy to vaccine components.
10. Individuals participating in any clinical trial with another investigational product 30 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
11. Individuals who have previously received any vaccines against typhoid fever (either oral live attenuated or injectable vaccines).
12. Individuals who received any other vaccines within 4 weeks prior to enrolment in this study or who are planning to receive any vaccine within 4 weeks from the study vaccine.
13. Individuals who have received blood, blood products and/or plasma derivatives including parenteral immunoglobulin preparations in the past 12 weeks.
14. Individuals who are part of study personnel or close family members to the personnel conducting this study.
15. Individuals with body temperature > 38.0 degrees Celsius within 3 days of intended study immunization.
16. BMI > 35 kg/m2.
17. Individuals with history of substance or alcohol abuse within the past 2 years.
18. Women who are pregnant or breast-feeding or of childbearing age who have not used any birth control measure one month prior to study start or do not plan to use acceptable birth control measures, for the duration of the study.
19. Females with history of stillbirth, neonatal loss, or previous infant with anomaly.
20. Individuals who have a previously ascertained or suspected disease caused by S. Typhi.
21. Individuals who have had household contact with/and or intimate exposure to an individual with laboratory confirmed S. Typhi.
22. Any condition which, in the opinion of the investigator may interfere with the evaluation of the study objectives.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for the Evaluation of Vaccination (CEV), Antwerp, Wilrijk (Antwerp), Belgium

REFERENCES:
- [Result] van Damme P, Kafeja F, Anemona A, Basile V, Hilbert AK, De Coster I, Rondini S, Micoli F, Qasim Khan RM, Marchetti E, Di Cioccio V, Saul A, Martin LB, Podda A. Safety, immunogenicity and dose ranging of a new Vi-CRM(1)(9)(7) conjugate vaccine against typhoid fever: randomized clinical testing in healthy adults. PLoS One. 2011;6(9):e25398. doi: 10.1371/journal.pone.0025398. Epub 2011 Sep 30. PMID 21980445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrollment: 04 OCT 10 Date of last visit: 18 NOV 10
Groups:
- NVGH Vi-CRM197 12.5 Mcg: 1 dose of 0.5 mL containing 12.5 mcg of Vi-CRM
- NVGH Vi-CRM197 5.0 Mcg: 1 dose of 0.5 mL containing 5.0 mcg of Vi-CRM
- NVGH Vi-CRM197 1.25 Mcg: 1 dose of 0.5 mL containing 1.25 mcg of Vi-CRM
- Typherix: 1 dose of 0.5 mL containing 25 mcg of Vi-PS
Period: Overall Study
Arm/Group | NVGH Vi-CRM197 12.5 Mcg | NVGH Vi-CRM197 5.0 Mcg | NVGH Vi-CRM197 1.25 Mcg | Typherix
Started | 22 | 22 | 22 | 22
Completed | 21 | 22 | 22 | 21
Not Completed | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVGH Vi-CRM197 12.5 Mcg | NVGH Vi-CRM197 5.0 Mcg | NVGH Vi-CRM197 1.25 Mcg | Typherix | Total
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 22 | 22 | 88
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (4.9) | 24.3 (5.4) | 24.0 (5.7) | 23.8 (5.5) | 24.1 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 17 | 15 | 61
  Male | 8 | 7 | 5 | 7 | 27
Region of Enrollment [Number; unit: participants]
  Belgium | 22 | 22 | 22 | 22 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any Post Immunization Reactions
Description: Solicited reactions collected during the 7-day period after vaccination are pain, erythema, induration, chills, malaise, myalgia, headache, arthralgia and fatigue
Time Frame: During the 7-day period after vaccination
Measure: Number; unit: participants
Arm/Group | NVGH Vi-CRM197 12.5 Mcg | NVGH Vi-CRM197 5.0 Mcg | NVGH Vi-CRM197 1.25 Mcg | Typherix
Number analyzed (Participants) | 21 | 22 | 22 | 22
participants | 18 | 19 | 22 | 16

2. Primary Outcome: Number of Subjects Reporting Adverse Events
Time Frame: During the 28-day period after vaccination
Measure: Number; unit: participants
Arm/Group | NVGH Vi-CRM197 12.5 Mcg | NVGH Vi-CRM197 5.0 Mcg | NVGH Vi-CRM197 1.25 Mcg | Typherix
Number analyzed (Participants) | 21 | 22 | 22 | 22
participants | 11 | 16 | 18 | 15

3. Primary Outcome: Anti-Vi ELISA (Enzyme Linked Immunosorbent Assay) Geometric Mean Concentration (GMC)
Time Frame: At 28 days after vaccination
Measure: Mean (95% Confidence Interval); unit: GMC
Arm/Group | NVGH Vi-CRM197 12.5 Mcg | NVGH Vi-CRM197 5.0 Mcg | NVGH Vi-CRM197 1.25 Mcg | Typherix
Number analyzed (Participants) | 21 | 21 | 19 | 20
GMC | 192 [129 to 286] | 111 [75 to 165] | 63 [41 to 95] | 37 [24 to 55]

4. Primary Outcome: Percentage of Subjects With at Least 4-fold Increase in Anti-Vi ELISA Titer
Time Frame: At 28 days after vaccination
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | NVGH Vi-CRM197 12.5 Mcg | NVGH Vi-CRM197 5.0 Mcg | NVGH Vi-CRM197 1.25 Mcg | Typherix
Number analyzed (Participants) | 21 | 21 | 19 | 20
percentage of subjects | 100 [84 to 100] | 100 [84 to 100] | 95 [74 to 100] | 95 [75 to 100]

ADVERSE EVENTS:
Arm/Group | NVGH Vi-CRM197 12.5 Mcg | NVGH Vi-CRM197 5.0 Mcg | NVGH Vi-CRM197 1.25 Mcg | Typherix
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 19/21 | 19/22 | 22/22 | 19/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVGH Vi-CRM197 12.5 Mcg (N=21) | NVGH Vi-CRM197 5.0 Mcg (N=22) | NVGH Vi-CRM197 1.25 Mcg (N=22) | Typherix (N=22)
diarrhoea (Gastrointestinal disorders) | 1 | 3 | 5 | 1
nausea (Gastrointestinal disorders) | 0 | 4 | 2 | 0
chills (General disorders) | 1 | 2 | 2 | 2
Fatigue (General disorders) | 7 | 11 | 8 | 7
injection site erythema (General disorders) | 3 | 2 | 2 | 0
injection site induration (General disorders) | 3 | 4 | 3 | 2
injection site pain (General disorders) | 17 | 16 | 21 | 9
malaise (General disorders) | 4 | 4 | 5 | 4
nasopharingitis (Infections and infestations) | 4 | 9 | 5 | 5
viral URTI (Infections and infestations) | 2 | 0 | 0 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4 | 3
headache (Nervous system disorders) | 11 | 11 | 12 | 10
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event that no publication of the Study results has been made by NVGH within twelve (12) months of Study database lock and no proposed publication is under discussion by the publication committee, Principal Investigator may publish its own Study results.